CLINICAL TRIAL: NCT05167994
Title: Preoperative Intensity-modulated Radiotherapy (IMRT) With Concurrent Anlotinib Hydrochloride for Localised Extremity or Trunk Sarcoma
Brief Title: Preoperative IMRT With Concurrent Anlotinib for Localised Extremity or Trunk Sarcoma （SPARE-01）
Acronym: SPARE-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, NINGNING LU, Principle Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2333
Record Dates: First submitted 2021-12-02; First posted 2021-12-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Sarcoma,Soft Tissue; Extremity; Trunk; Anlotinib; Intensity-modulated Radiotherapy; Major Wound Complications
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib arm (Experimental): Pre-operative IMRT with concurrent and sequential Anlotinib
  Interventions: Drug: Anlotinib hydrochloride

INTERVENTIONS:
Drug: Anlotinib hydrochloride — Anlotinib 12mgQD, from D1 of pre-operative IMRT to 1 month after end of IMRT

SUMMARY:
To investigate the safety and efficacy of preoperative IMRT and concurrent Anlotinib Hydrochloride for primary truncal or extremity soft tissue sarcoma; To investigate the Quality of life and extremity function post-combination treatment; To study the mechanism of radio-sensitizing effects of Anlotinib Hydrochloride for primary truncal or extremity soft tissue sarcoma; To assess the relationship between the MRI imaging, pathological findings and local control.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18-yo
* Histology proven soft tissue sarcoma of truncal or extremity, deemed appropriate for preoperative radiotherapy and conservative surgery by multidisciplinary discussion.
* ECOG 0-3
* Histology reviewed by reference pathologist
* Lesion can be assessed
* Can tolerate radiotherapy and Anlotinib
* Agree contraception.
* Informed consent: All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed

Exclusion Criteria:

* No gross tumor post-resection in other center.
* Contraindications to Anlotinib, including allergic to Anlotinb, active bleeding, ulcer, enteric perforation, enteric obstruction, uncontrolled hypertension, Grade 3 to 4 cardiac insufficiency (per NYHA criteria), and severe hepatic or renal insufficiency (Grade 4), etc.
* Dermatofibrosarcoma protuberans(DFSP), Desmoids, etc.
* Benign histology
* Secondary cancer within 5 years (except cervical carcinoma in situ or early-stage skin basal cell carcinoma)
* STS can be cured by extensive operation alone.
* Previous irradiation to the same area
* Radiological evidence of distant metastases
* Other contraindications, can't tolerate operation or other treatment needed in this study.
* Neoadjuvant chemotherapy given or planned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Major wound complications | 4-months post-surgery

SECONDARY OUTCOMES:
Acute and late toxicities | acute toxicities were evaluated during and 3 months after IMRT, late toxicities were evaluted after 6 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Quality of Life | pre-IMRT, end of IMRT, 1 months post-IMRT, and every 3 to 6 months during follow-up
  Evaluate quality of life by QOL questionnaires at different time points
Extremity function | pre-IMRT, end of IMRT, 1 months post-IMRT, and every 3 to 6 months during follow-up
  Evaluate quality of life by MSTS forms at different time points
Pathological remission rate | 2 weeks after operation
  evaluate the tumor remission rate microscopically
Local control | 2-year
Overall Survival | 2-year

CONTACTS AND LOCATIONS:
Locations (1):
- Radiotherapy Department of Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China